CLINICAL TRIAL: NCT06498258
Title: The Effect of Positive Psychotherapy Balance Model Based Psychoeducation on Balanced Life, Psychological Well-Being and Self-Efficacy in Caregivers of Oncology Patients.
Brief Title: Positive Psychotherapy Balance Model Based Psychoeducation for Caregivers of Oncology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Servet CİHAN (Other)
Responsible Party: Sponsor-Investigator, Servet CİHAN, Eğitim hemşiresi, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ServetCİHANCEmilTascıoğluERHO
Record Dates: First submitted 2024-06-25; First posted 2024-07-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Kolon Kanseri
Keywords: pozitif psikoterapi; Kanser; psikolojik refah; öz yeterlilik; yaşam dengesi

STUDY DESIGN:
Intervention Model Description: In this study, positive psychotherapy balance model applied to individuals caring for oncology patients the effect of psychoeducation intervention on balanced life, psychological well-being and self-efficacy. It will be carried out as a randomised control group experimental research with pretest-posttest follow-up.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deneysel grup (Experimental): positive psychotherapy balance model based psychoeducation intervention
  Interventions: Other: Pozitif Psikoterapi Denge Modeli Temelli Psikoeğitim
- kontrol grubu (No Intervention): positive psychotherapy balance model TRAINING

INTERVENTIONS:
Other: Pozitif Psikoterapi Denge Modeli Temelli Psikoeğitim — In this study, it can be said that adopting a loving, connected and balanced state of mind in the face of the difficulties experienced and responsibilities undertaken by caregivers will increase the joy, meaning and self-sufficiency in life and as a result, it can positively contribute to their level of well-being. All these results are important for caregivers to be able to recognise their own resources, to maintain their life balance, to develop a positive perspective towards themselves, to make subjective evaluations and to recognise their strengths.
  Arms: deneysel grup

SUMMARY:
In this study, positive psychotherapy balance model applied to individuals caring for oncology patients the effect of psychoeducation intervention on balanced life, psychological well-being and self-efficacy. It will be carried out as a randomised control group experimental research with pretest-posttest follow-up. The independent variable of the study is positive psychotherapy balance model based psychoeducation intervention. The dependent variables are Balanced Life Scale, Psychological Well-Being Scale, Self-Efficacy Scale. The control variables are the socio-demographic characteristics of the participants (gender, age, educational status, marital status, etc.) and the characteristics related to the caregiving process (duration of care, time allocated for care, etc.).

Hypothesis 1: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of balanced life.

H1.1: Positive psychotherapy balance model based psychoeducation has an effect on increasing the level of success.

H1.2: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of relationship.

H1.3: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of future/meaning/spirituality.

H1.4: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the body level.

Hypothesis 2: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of psychological well-being.

Hypothesis 3: Positive psychotherapy balance model based psychoeducation has an effect on increasing general self-efficacy level.

Research data will be collected with data collection tools after obtaining ethics committee and institutional permission. Psychoeducation based on the positive psychotherapy balance model will be carried out face-to-face with caregivers of individuals with colorectal cancer in a city hospital.

The population of the study will consist of caregivers of individuals diagnosed with colorectal cancer in a city hospital. The sample of the study was calculated by performing power analysis with GPower 3.1.9.4 programme. As a result of the power analysis based on a similar study for the research designed as a control and an intervention group, the total sample size was calculated as 38 people in the groups of 19 people at the 85% Power 0.05 alpha significance level, with the prediction that the difference in the medium effect size f=0.25 between the groups in the pre and post evaluations for the two groups would be considered statistically significant. Considering the possibility of caregivers dropping out or being excluded from the study, it was decided to include 8 additional people, 4 in each group. A total of 46 caregivers in the intervention and control groups will constitute the sample of the study.

Which caregivers will be in the intervention group and which will be in the control group will be determined according to the randomisation table determined via the internet https://www.randomizer.org/. Group 1: Intervention Group, Group 2: Control Group. Afterwards, they will be assigned to the groups in accordance with the order in the randomisation table. The randomisation result will be indicated in the form of a table.

Personal information form, Balanced Life Scale, Psychological Well-Being Scale and Self-Efficacy Scale will be used as data collection tools.

Data collection tools will be applied to all caregivers who agree to participate in the study and meet the inclusion criteria, and a brief information about the psychoeducation process will be given. Psychoeducation based on Positive Psychotherapy Balance Model will be conducted in 5 sessions (5 weeks), one day a week, 90-120 minutes. The control group will receive a one-session (60 minutes) information training after 3 weeks.

After all sessions are completed, post-tests will be applied to the intervention group and the control group.. Follow-up data will be collected from the intervention and control groups 3 months after the psychoeducation programme is completed. After the end of the study, PPT Balance Model Based Psychoeducation will be given to the caregivers in the control group.

DETAILED DESCRIPTION:
İntroduction and Objective: Cancer is one of the leading chronic health problems in terms of mortality and morbidity all over the world, accompanied by many symptoms, requiring a long-term treatment process, and requiring attentive care not only in the hospital but also in the home environment. For an individual with a diagnosis of cancer, the caregiver is involved in all physical, emotional, social, spiritual and economic dimensions of patient care. Caregivers are involved in the they play an important role in the care, adaptation and management of the disease. Struggling with a vital disease such as cancer is a serious physical, economic and social challenge not only for the patient but also for the patients family and close environment, especially in terms of mental health status affects in a sense. The continuous and intensive nature of caregiving, combined with other responsibilities in the life spheres of individuals caring for oncology patients, turns into a dependent, unidirectional, intensive and long-term obligation that disrupts the care-giving-caregiving relationship, distresses the caregivers life, and creates a conflict between the care roles of the caregiver with family relationships, entertainment, work and social life roles. Caregivers need to find a balance to resolve the conflict between the responsibilities of the care role and their own needs and demands. However, they benefit from limited training, information and support in the caregiving role.

The principle of balance, which is one of the principles of positive psychotherapy, argues that it is possible for individuals to cope with their conflicts by allocating their life energies to four areas in a balanced way. In accordance with the principle of balance, individuals should use the areas of body, relationship, success and future/spirituality in a balanced way in order to solve the problems they experience. Because, according to positive psychotherapy, it is possible for individuals to have a fully healthy and productive life with the importance they will give to these four basic life dimensions and the balanced use of the time and energy they will spend. In the context of positive psychotherapy, an individual who has a balanced life goal and also has high general self-efficacy skills is expected to be more courageous and willing to show the necessary efforts to maintain a balanced life. Because the individual with high general self-efficacy skills will have a strong belief in overcoming the problems he/she may encounter despite the effort he/she will make for a balanced life, and thus, the individual who has the desire to live a balanced life and can find the competence to make the necessary efforts will be able to keep his/her motivation high to continue his/her efforts as he/she sees the positive changes in his/her life with the steps he/she will take. The concept of psychological well-being, which focuses on the self-development and growth of the individual by realising his/her own meaning, competence and capacity based on the individuals own self-powers and competencies, is the natural result of the process experienced by the individual aiming for such a life at this point. In this direction, it can be said that adopting a loving, connected and balanced state of mind in the face of the difficulties experienced by caregivers and the responsibilities they undertake will increase the joy, meaning, self-sufficiency in life and, as a result, may contribute positively to their level of well-being. All these results help caregivers to recognise their own resources, maintain their life balance, and adopt a positive perspective towards themselves.

Materials and Methods: In this study, positive psychotherapy balance model applied to individuals caring for oncology patients the effect of psychoeducation intervention on balanced life, psychological well-being and self-efficacy. It will be carried out as a randomised control group experimental research with pretest-posttest follow-up. The independent variable of the study is positive psychotherapy balance model based psychoeducation intervention. The dependent variables are Balanced Life Scale, Psychological Well-Being Scale, Self-Efficacy Scale. The control variables are the socio-demographic characteristics of the participants (gender, age, educational status, marital status, etc.) and the characteristics related to the caregiving process (duration of care, time allocated for care, etc.).

Hypothesis 1: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of balanced life.

H1.1: Positive psychotherapy balance model based psychoeducation has an effect on increasing the level of success.

H1.2: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of relationship.

H1.3: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of future/meaning/spirituality.

H1.4: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the body level.

Hypothesis 2: Positive psychotherapy balance model-based psychoeducation has an effect on increasing the level of psychological well-being.

Hypothesis 3: Positive psychotherapy balance model based psychoeducation has an effect on increasing general self-efficacy level.

Research data will be collected with data collection tools after obtaining ethics committee and institutional permission. Psychoeducation based on the positive psychotherapy balance model will be carried out face-to-face with caregivers of individuals with colorectal cancer in a city hospital.

The population of the study will consist of caregivers of individuals diagnosed with colorectal cancer in a city hospital. The sample of the study was calculated by performing power analysis with GPower 3.1.9.4 programme. As a result of the power analysis based on a similar study for the research designed as a control and an intervention group, the total sample size was calculated as 38 people in the groups of 19 people at the 85% Power 0.05 alpha significance level, with the prediction that the difference in the medium effect size f=0.25 between the groups in the pre and post evaluations for the two groups would be considered statistically significant. Considering the possibility of caregivers dropping out or being excluded from the study, it was decided to include 8 additional people, 4 in each group. A total of 46 caregivers in the intervention and control groups will constitute the sample of the study.

Which caregivers will be in the intervention group and which will be in the control group will be determined according to the randomisation table determined via the internet. Group 1: Intervention Group, Group 2: Control Group. Afterwards, they will be assigned to the groups in accordance with the order in the randomisation table. The randomisation result will be indicated in the form of a table.

Personal information form, Balanced Life Scale, Psychological Well-Being Scale and Self-Efficacy Scale will be used as data collection tools.

Data collection tools will be applied to all caregivers who agree to participate in the study and meet the inclusion criteria, and a brief information about the psychoeducation process will be given. Psychoeducation based on Positive Psychotherapy Balance Model will be conducted in 5 sessions (5 weeks), one day a week, 90-120 minutes. The control group will receive a one-session (60 minutes) information training after 3 weeks.

After all sessions are completed, post-tests will be applied to the intervention group and the control group.. Follow-up data will be collected from the intervention and control groups 3 months after the psychoeducation programme is completed. After the end of the study, PPT Balance Model Based Psychoeducation will be given to the caregivers in the control group.

Ethics committee and institutional permission will be obtained from Istanbul Prof. Dr. Cemil Taşcıoğlu City Hospital Interventional Health Sciences Research Ethics Committee for the implementation of the research. After the individuals included in the study are informed about the research, their written and verbal consent will be obtained through data collection forms.

SPSS 15.0 for Windows programme will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* To be in the age group of 18 and above
* To have a score of 90 and below on the Barthel VAS Index
* To be at least primary school graduate
* To have no psychiatric illness (diagnosis)
* To have no communication and comprehension disability related to vision, hearing
* To live in Istanbul

Exclusion Criteria:

* Not having attended all sessions of the training programme
* Not having answered any of the pre-test, post-test and follow-up tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Balanced life levels will be measured using the Balanced Life Scale with psychoeducation based on the positive psychotherapy balance model for individuals caring for oncology patients. | 5 hafta
  Balanced life levels will be measured using the Balanced Life Scale with psychoeducation based on the positive psychotherapy balance model for individuals caring for oncology patients. (Face-to-face training will be given)
Psychoeducation based on the positive psychotherapy balance model will be provided to individuals caring for oncology patients and their general self-efficacy levels will be measured using the General Self-Efficacy scale. | 5 hafta
  Psychoeducation based on the positive psychotherapy balance model will be provided to individuals caring for oncology patients and their general self-efficacy levels will be measured using the General Self-Efficacy scale. (Face-to-face training will be given)
Psychological well-being levels will be measured using the Psychological Well-Being Scale with psychoeducation based on the positive psychotherapy balance model for individuals caring for oncology patients. | 5 hafta
  Psychological well-being levels will be measured using the Psychological Well-Being Scale with psychoeducation based on the positive psychotherapy balance model for individuals caring for oncology patients. (Face-to-face training will be given)

CONTACTS AND LOCATIONS:
Overall Officials: Servet Cihan, Principal Investigator — Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Kağithane, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] undefined